CLINICAL TRIAL: NCT00484172
Title: Genomic Search for Childhood Obesity Genes-A Pilot Study
Status: Withdrawn | Type: Observational
Why Stopped: Study Withdrawn due to Investigator leaving
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 07 03-045E
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: blood draws

SUMMARY:
The purpose of this study is to screen a pediatric population (ages 2-8) for genes associated with childhood obesity.

DETAILED DESCRIPTION:
The incidence of childhood obesity has been growing at an epidemic rate for the past several years, in part due to the lack of understanding of mechanisms at a molecular level. This study will screen a healthy general pediatric population age 2 to 8 for potential genes associated with childhood obesity using whole genomic gene arrays. Patients with BMI values equal to or greater than the 85th percentile will be compared to patients with a BMI below or equal to the 15th percentile. The INSIG2 gene will be specifically studied because of its identification in several populations of obese subjects. The differences in gene expression of the 2 groups will then be used to identify new genes for investigation in childhood obesity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2-8, predominately Caucasian to minimize population stratification

Exclusion Criteria:

* Chronic diseases (diabetes, cancer, etc) and known syndromes

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 2-8 years old
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merlin G Butler, M.D., Ph.D., Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States